CLINICAL TRIAL: NCT06227533
Title: Comparison Between Two Regenerative Scaffolds Outcome in The Treatment of Mature Teeth With Necrotic Pulp and Periapical Radiolucency
Brief Title: Comparison Between Two Regenerative Scaffolds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Taghreed Salah, lecturer assistant, Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENDOD-104-1-E
Record Dates: First submitted 2024-01-16; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Pulp Necroses
Keywords: regeneration, mature teeth
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Intervention Model Description: The current study was designed as randomized controlled clinical trial with an allocation ratio 1:1
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Eighteen papers were numbered from 1 to 18 and individually packed in opaque envelopes. Each patient picked an envelope before the beginning of the second visit. The number in the envelope determined the regenerative protocol which was to be performed for the participant. The patient was not informed of what procedure he/she was subjected to
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF group (Experimental): Five ml blood will be drawn from the patient's right median cubital vein into a test tube without the addition of an anticoagulant and centrifuged immediately at 3000 rpm for 10 minutes
  Interventions: Procedure: Endodontic regeneration using concentrated growth factor compared with Platelet rich fibrin
- CGF group (Experimental): Ten ml of intravenous blood sample from the patient will be obtained and placed in centrifuge tubes without anticoagulants; accelerated for 30 seconds; centrifuged at 2700 rpm for 2 min, 2400 rpm for 4 min, 2700 rpm for 4 min, and 3000 rpm for 3 min; and decelerated for 36 secs to stop
  Interventions: Procedure: Endodontic regeneration using concentrated growth factor compared with Platelet rich fibrin

INTERVENTIONS:
Procedure: Endodontic regeneration using concentrated growth factor compared with Platelet rich fibrin — regeneration of mature necrotic teeth with periapical abscess using concentrated growth factor compared with Platelet rich fibrin to allow healing of periapical lesion and regaining sensibility
  Other Names: Endodontic regeneration of mature teeth

SUMMARY:
This study was performed to compare endodontic regeneration outcome in necrotic mature single rooted teeth with periapical radiolucency using platelet rich fibrin (PRF) & concentrated growth factor (CGF) as a different natural scaffold by evaluation of:

* Regaining pulp sensibility by thermal test (hot and cold)
* Periapical healing using digital radiography and selected samples will be evaluated using Cone Beam Computed Tomography (CBCT).

DETAILED DESCRIPTION:
The current study was designed as randomized controlled clinical trial with an allocation ratio 1:1 and conducted in the clinic of Endodontic Department, Faculty of Dental Medicine for Girls, Al-Azhar University. The study was designed, analyzed and interpreted according to the Consolidated Standards of Reporting Trials (CONSORT 2010) checklist of information. Ethical approval for the human research was obtained in accordance with guidelines from Research Ethics Committee (REC) of the institute with the code number: P-EN-21-02. All patients read and signed an informed consent form with details about the study along with the benefits and risks of the therapy (Appendix A).A total of thirty-six patients were examined for this study.

After clinical and radiographic examinations only eighteen patients from cases that were fulfilling the inclusion criteria were selected according to sample size calculation. Eighteen cases was divided randomly into two groups (9 cases each):

Group I (PRF group):

Preparation of PRF:

Five ml blood was drawn from the patient's right median cubital vein into a test tube without the addition of an anticoagulant and centrifuged immediately at 3000 rpm for 10 minutes

Group II (CGF group):

Preparation of CGF:

Ten ml of intravenous blood sample from the patient will be obtained and placed in centrifuge tubes without anticoagulants; accelerated for 30 seconds; centrifuged at 2700 rpm for 2 min, 2400 rpm for 4 min, 2700 rpm for 4 min, and 3000 rpm for 3 min; and decelerated for 36 secs to stop.

Methodology:

Common treatment protocol will be as follow:

First visit: tooth was isolated using rubber dam followed by access cavity preparation and working length determination. Mechanical preparation of root canal was performed using rotary instrumentation then the canal was irrigated by 1.5% NaOCl between each successive file. After drying the canal with paper point, Calcium hydroxide as intracanal medicament was placed. The access cavity was sealed with a cotton pellet and glass ionomer cement for three weeks.

Second visit: plain anesthesia without a vasoconstrictor was administrated. Glass ionomer was removed under the isolation with rubber dam. Calcium hydroxide was flushed from the canal using 5ml sterile saline followed by irrigation using 20ml of 17% ethylene diamine tetra acetic acid (EDTA) then drying the canal using paper point. Intentional over-instrumentation 3 mm beyond the apex was done using sterile #35 k file to induce bleeding inside the canal followed by placement of PRF and CGF inside the canal in group I and group II respectively followed by placement of 3 mm mineral trioxide aggregate (MTA) below cementoenamel junction and the coronal cavity will be sealed using composite.

The regeneration outcome will be evaluated 6 month and 1 year follow up, clinically using thermal test to ensure the restoration of pulp sensibility or not and radiographically using digital radiograph to assess the periapical healing. Selected samples will be evaluated using Cone Beam Computed Tomography (CBCT).

ELIGIBILITY:
Inclusion Criteria:

* Agree to participate in this study and provide informed consent
* Age range of 18 - 30 years
* Free from systemic diseases.
* Having necrotic single-rooted maxillary central incisor with mature root and periapical radiolucency sized up to 5mm.
* Restorable teeth that can be isolated with rubber dam and restored with direct coronal restoration.

Exclusion Criteria:

* Pregnant females.
* Generalized chronic periodontitis.
* Non-restorable teeth.
* Previous root canal treatment.
* Developmental anomalies.
* External and / or internal root resorption.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
healing | 1 year
  The elimination of symptoms and the evidence of periapical bony healing assessed radiographically (incidence of bone formation at the apex of root which indicate complete healing of chronic periapical abscess which assessed by periapical radiograph and cbct at 6 months & 1 year after treatment , as it appear radiolucency in radiograph which decrease by time that indicate complete healing of abscess and reformation of bone apically

SECONDARY OUTCOMES:
regaining of pulp sensibility | 1 year
  restoration of normal pulp sensation assessed by thermal test (hot using hot water in plastic syringe & cold using endo ice ) after isolation of the tooth.. thermal test was done before treatment then 6 month &1 year follow up and ask the patient about his sensation

CONTACTS AND LOCATIONS:
Overall Officials: heba abd el kafy, lecturer, Study Director — faculty of dental medicine for girls Al Azhar University
Locations (1):
- faculty of dental medicine for girls Al Azhar University, Cairo, Egypt

REFERENCES:
- [Derived] Salah T, Hussein W, Abdelkafy H. Regenerative potential of concentrated growth factor compared to platelet-rich fibrin in treatment of necrotic mature teeth: a randomized clinical trial. BDJ Open. 2025 Feb 3;11(1):10. doi: 10.1038/s41405-024-00288-3. PMID 39900647